CLINICAL TRIAL: NCT02931162
Title: Efficacy of Moxibustion Treatment on Patients With Ulcerative Colitis
Brief Title: The Effects of Moxibustion on Ulcerative Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Institute of Acupuncture, Moxibustion and Meridian (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UC-Brain
Record Dates: First submitted 2016-09-25; First posted 2016-10-12 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2018-06

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Herb-partitioned moxibustion (Experimental): Drug: Herbal cake, Device: Moxibustion. Herbal cakes formula: Monkshood 10g, Cinnamon 2g, Salvia miltiorrhiza 3g, Flos Carthami 3g, Radix Aucklandiae 2g. Herbs are smashed into powder. Every 2.5g medicine powder is mixed with 3g millet wine and then pressed into herbal cakes using a specific mold. Each cake should be 23mm in diameter and 5mm in height. Then, ignited moxa cones are placed on top of each herbal cake. Herbal cakes with moxa cones will be positioned at acupuncture points ST25 and ST37. The entire treatment will be done once a day for 1 moxa cone every acupuncture point, 30 minutes at a time, 3 times a week, for a total of 12 weeks.
  Interventions: Other: Herb-partitioned moxibustion
- Sham herb-partitioned moxibustion (Sham Comparator): Drug: Herbal cake, Device: Sham moxibustion. Herbal cakes formula: Monkshood 10g, Cinnamon 2g, Salvia miltiorrhiza 3g, Flos Carthami 3g, Radix Aucklandiae 2g. Herbs are smashed into powder. Every 2.5g medicine powder is mixed with 3g millet wine and then pressed into herbal cakes using a specific mold. Each cake should be 23mm in diameter and 5mm in height. Then, ignited moxa cones are placed on top of each herbal cake. Small cardboard sheets with the same size as the herbal cakes will be wrapped with aluminum foil and placed under each herbal cake. These herbal cakes will be positioned at acupuncture points ST25 and ST37. The entire treatment will be done once a day for 1 moxa cone every acupuncture point, 30 minutes at a time, 3 times a week, for a total of 12 weeks.
  Interventions: Other: Sham herb-partitioned moxibustion

INTERVENTIONS:
Other: Herb-partitioned moxibustion — Patients receive herb-partition moxibustion 3 times a week, once a day for 30 minutes, for a total of 12 weeks.
  Other Names: Treatment Group
  Arms: Herb-partitioned moxibustion
Other: Sham herb-partitioned moxibustion — Patients receive sham herb-partition moxibustion 3 times a week, once a day for 30 minutes, for a total of 12 weeks.
  Other Names: Control Group
  Arms: Sham herb-partitioned moxibustion

SUMMARY:
To investigate the mechanism and effects of moxibustion on patients with ulcerative colitis.

DETAILED DESCRIPTION:
A total of 60 patients with UC were randomly divided into the following 2 groups: a) Herb-partition moxibustion (Treatment Group) and b) Sham herb-partition moxibustion (Control Group). All patients in the trial will be treated with moxibustion 3 times a week, once a day for 30 minutes, for a total of 12 weeks. MRI will be used to observe the changes on brain structure and function in patients with UC, and further research on the characteristics of the brain nerve response of these patients with herb-partition moxibustion. In addition, tissue morphology and molecular biology tests will be conducted to observe the regulation and expression of VDR and antimicrobial peptides in the intestinal mucosa of UC patients. All these steps will be done in order to provide experimental basis for the mechanism of the effects of herb-partition moxibustion in the treatment of UC.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnosis of UC
* Mayo ≤10
* Patients do not receive any medicine, or if they are receiving medicine, it should be aminosalicylates and/or prednisone (dose ≤15mg and have taken at least 1 month), and must kept the same dose as before throughout the trial;
* Patients should have not received antibiotic, biologicals within 3 months prior to entering the study;
* Signing a written informed consent.

Exclusion Criteria:

* Patients with cardiac, encephalic, hepatic, nephric, hematopoietic system, psychotic or any other serious diseases;
* Pregnancy or lactation;
* The psychiatric patients;
* Current or prior history of neurosurgery, head injury, cerebrovascular insult, or brain trauma involving loss of consciousness;
* Learning disability;
* Claustrophobia;
* Presence of metallic implants in the body;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-08-23 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Mayo score | 3 months
  Assay for the ulcerative colitis desease activity index. It is constructed by four scales, Including stool frequency、rectal bleeding、mucosal appearance at endoscopy and physician rating of disease activity. Every scale can be scored with o ,1 ,2 or 3 according to the activity index of scale. Scores should be compared to previous scores taken for a patient. The higher the score (minimum 0 point and maximum 12 points), the more severe the ulcerative colitis.

SECONDARY OUTCOMES:
MRI | 3 months
  Brain structure(gray matter, white matter structures) changes examined by MRI
functional MRI | 3 months
  Brain resting state activity changes examined by functional MRI
mucosal pathology; Baron score; | 3 months
  using electronic colonoscopy
Inflammatory Bowel Disease Questionnaire(IBDQ) | 3 months
  Life quality was determined by the total score of the 32 questions. Each question is given 1-7 different degrees of answer. One represents the heaviest degree and seven represents the lightest degree. The lower the score (minimum 32 points and maximum 224 points), the worse the life quality.
Laboratory tests for disease activity: C-reaction protein | 3 months
  Assay for the quantification of total C-reaction protein in serum.(Normal reference value:<10mg/L)
Laboratory tests for disease activity: Erythrocyte sedimentation rate | 3 months
  Assay for the quantification of total Erythrocyte sedimentation rate in serum.(Normal reference value: male 0～15mm/h; female 0～20mm/h)
The serum concentrations of 1,25-dihydroxyvitamin D3 | 3 months
  The serum levels of 25(OH)D concentration.
symptom score | 3 months
  Observe the abdominal pain, bloody stool, intolerance of cold, soreness and weakness of waist an knees, diarrhea, mucous stool, tenesmus, anorexia and lassitude score.
Visual Analogue Scale(VAS) | 3 months
  Obserb the degree of abdominal pain and ventosity. Draw a 10 cm horizontal line on the paper, one end of which is 0, indicating no pain; The other end is 10, which means pain; The middle part indicates different degrees of pain. Ask the patient to make a mark on the line to indicate the degree of pain based on how he or she feels. The mean value of mild pain was 2.57 + / - 1.04. The mean of moderate pain was 5.18 + / - 1.41. The mean value of severe pain was 8.41 + / - 1.35 .
Hospital Anxiety and Depression Scale(HADS) | 3 months
  The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 .The higher the total score (minimum 0 point and maximum 21 points), the more severe the anxiety or depression
Self-Rating Anxiety Scale(SAS) | 3 months
  The SAS is a 20-item self-report assessment device built to measure anxiety levels. Each question is scored on a Likert-type scale of 1-4 (based on these replies: "a little of the time," "some of the time," "good part of the time," "most of the time").The total raw scores range from 20-80.The raw score then needs to be converted to an "Anxiety Index" score using the chart on the paper version of the test that can be found on the link below. The "Anxiety Index" score can then be used on this scale below to determine the clinical interpretation of one's level of anxiety:
  20-44 Normal Range 45-59 Mild to Moderate Anxiety Levels 60-74 Marked to Severe Anxiety Levels 75 and above Extreme Anxiety Levels
Self-rating Depression Scale(SDS) | 3 months
  The SDS is a 20-item self-report assessment device built to measure depression levels. Each question is scored on a Likert-type scale of 1-4 (based on these replies: "a little of the time," "some of the time," "good part of the time," "most of the time").The total raw scores range from 20-80.The raw score then needs to be converted to an "Depression Index" score using the chart on the paper version of the test that can be found on the link below. The "Depression Index" score can then be used on this scale below to determine the clinical interpretation of one's level of anxiety:
  20-44 Normal Range 45-59 Mild to Moderate Depression Levels 60-74 Marked to Severe Depression Levels 75 and above Extreme Depression Levels
The serum levels of IL-12/23 p40 | 3 months
  The changes of serum IL-12/23 p40 concentration before and after treatment were observed.
The expression of Cyp27b1, Reg IV and VDR mRNA in mucosa | 3 months
  The relative quantity of Cytochrome p450 27B1(Cyp27b1), Reg IV and Vdr by real-time quantitative PCR.
The expression of Reg4 and VDR in mucosa | 3 months
  The protein expressions of Reg IV and VDR in UC colon mucosa were detected by immunohistochemistry.
The level of TNF-α, IFN-γ, IL-2 and LPS in plasma | 3 months
  The plasma lever of IL-2, LPS, IFN-γ and TNF-α by using ELISA method.
The expression of IL-12, TLR4, MyD88, IRAK, TRAF6 and NF-κB in mucosa | 3 months
  IL-12, TLR4, MyD88, IRAK, TRAF6 and NF-κB in UC colon mucosa were detected by immunohistochemistry.

OTHER OUTCOMES:
Safety Assessment | 3 months
  With Administration Events reports record the adverse reaction treatment process, with the moxibustion treatment of safety evaluation. Such as the incidence and severity of scald, skin allergic, vasodepressor syncope etc. Also record subjects's vital signs, consist of body temperature, blood pressure and pulse.

CONTACTS AND LOCATIONS:
Overall Officials: Huangan Wu, Doctor, Study Director — Shanghai Institute of Acupuncture-Moxibustion and Meridian, Shanghai University of Traditional Chinese Medicine.
Locations (1):
- Outpatient department of Shanghai Research Insititute of Acupuncture and Meridian, Shanghai, Xuhui, China

IPD SHARING:
Plan to Share IPD: Undecided